CLINICAL TRIAL: NCT03136835
Title: Maternal Hyperoxygenation in Congenital Heart Disease
Acronym: MATCH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mike Seed, Dr. Michael Seed, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000048468
Record Dates: First submitted 2015-10-28; First posted 2017-05-02 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot (Experimental): Maternal Hyperoxygenation (4L/min via nasal prongs)
  Interventions: Drug: Maternal Hyperoxygenation

INTERVENTIONS:
Drug: Maternal Hyperoxygenation — Oxygen via nasal prongs at up to 4L/min continuously during 2nd and 3rd trimester of pregnancy until birth
  Other Names: Oxygen

SUMMARY:
A pilot study investigating the safety and feasibility of chronic maternal hyperoxygenation in the setting of fetal congenital heart disease

DETAILED DESCRIPTION:
The aim of the study is to investigate the safety and feasibility of chronic maternal hyperoxygenation in pregnancies affected by fetal congenital heart disease, specifically those pregnancies in which the fetus has single ventricle physiology with aortic arch obstruction. The treatment has a potentially neuroprotective effect on the fetus. This would be desirable as the neurodevelopmental outcomes of the survivors of this form of congenital heart disease are significantly below normal. However, transplacental oxygen has not been tried in this setting, and so before embarking on a trial, the investigators need to establish that the treatment is safe and feasible. This will be accomplished by recruiting subjects which meet the eligibility criteria and commence treatment at the time of diagnosis, usually in the second trimester, and by comparing outcomes with a historical cohort with CHD diagnoses with no oxygen intervention. The oxygen will be delivered to the mother via nasal prongs continuously at a rate of up to 4 L/min. Oxygen concentrators will be supplied to the subjects' homes, and a range of portable devices will also be provided to allow them to continue with usual activities of daily living. A series of follow up appointments will be arranged to check the status of the mother and fetus. Mothers will be invited to keep a diary of their adherence to the treatment. A range of routine clinical and research data on the condition of the fetus and newborn will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Between 20-32 weeks gestation
* Diagnosis of fetus with a single ventricular ventricular heart
* Delivering at Mount Sinai Hospital
* Written informed consent

Exclusion Criteria:

* Opting for termination of pregnancy/ comfort care
* Normal exclusions for MRI (e.g. claustrophobia, cardiac pacemaker, etc.)
* BMI >37.0
* Infections/ anemia
* Smoker
* Serious cardiorespiratory co-morbidities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
The general condition of the child and mother at the time of birth | 2 years
  The general condition of the child and mother at birth, classified by any maternal or fetal adverse events. Adverse events will also be classified as mild, moderate, severe, life-threatening or disabling, or fatal. The investigators will further define adverse events in terms of their effect on usual daily activities as follows: mild (an awareness of symptoms but easily tolerated), moderate (symptoms interfere with normal daily activities) or severe (symptoms are incapacitating, with the inability to perform daily activities). As unexpected adverse effects are by definition difficult to predict, the investigators use a variety of sources of information to identify possible side effects of the treatment including participant diaries, direct observations, participant reports, laboratory reports and other medical reports.
The duration of oxygen therapy tolerated by the subjects | 2 years
  This will be as a proportion of the maximum potential duration if the subjects had adhered to the continuous therapy from enrollment to birth.
  If the treatment is not tolerable by a substantial number (e.g. >10%) of subjects for significant periods of time (e.g. more than 8 hours a day) in the pilot study then this will be considered a negative result, i.e. that the treatment is not feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Seed, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lee FT, Sun L, Szabo A, Milligan N, Saini A, Chetan D, Hunt JL, Macgowan CK, Freud L, Jaeggi E, Van Mieghem T, Kingdom J, Miller SP, Seed M. Safety and feasibility pilot study of continuous low-dose maternal supplemental oxygen in fetal single ventricle heart disease. Ultrasound Obstet Gynecol. 2024 Oct;64(4):493-503. doi: 10.1002/uog.27657. PMID 38629477